CLINICAL TRIAL: NCT03796650
Title: COmparative Effectiveness of IntestinaL MicrobiOta Versus VaNcomycin for Primary C. Difficile Infection - RandomiZEd Trials
Brief Title: Fecal Transplantation for Primary Clostridium Difficile Infection
Acronym: COLONIZE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Pre-specified non-inferiority criterion met at interim analysis.
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); University Hospital of North Norway (Other); Haukeland University Hospital (Other); Helse Nord-Trøndelag HF (Other); Vestre Viken Hospital Trust (Other); The Hospital of Vestfold (Other); Sykehuset Telemark (Other Government); Alesund Hospital (Other); University Hospital, Akershus (Other); Lovisenberg Diakonale Hospital (Other); Sorlandet Hospital HF (Other Government); Ostfold Hospital Trust (Other); Diakonhjemmet Hospital (Other); Nordlandssykehuset HF (Other); Sykehuset Innlandet HF (Other); Helse Stavanger HF (Other Government)
Responsible Party: Principal Investigator, Kjetil Garborg, Joint Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COLONIZE
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile; Intestinal microbiota therapy; Fecal microbiota transplantation; Investigator-initiated; Antibiotics; Diarrhea
MeSH Terms: conditions — Clostridium Infections; Diarrhea | interventions — Fecal Microbiota Transplantation; Vancomycin

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with two parallel treatment arms with a 1:1 allocation.
Who Masked: Outcomes Assessor
Masking Description: An open-label, partly assessor blinded trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fecal microbiota transplantation (Experimental): Fecal microbiota from healthy, screened stool donors at the University Hospital of North Norway. Patients will receive one FMT enema immediately after enrolment.
  Interventions: Other: Fecal microbiota transplantation
- Antibiotic treatment (Active Comparator): Patients randomized to the control group will receive a ten-day course of oral vancomycin four times a day. This is according to international guidelines for primary C. difficile treatment.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Other: Fecal microbiota transplantation — 50 g donor feces suspended in saline with added glycerol, administered by a enema kit.
  Other Names: FMT; IMT; Bacteriotherapy
  Arms: Fecal microbiota transplantation
Drug: Vancomycin — Peroral vancomycin 125 mg q.i.d. for ten days.
  Arms: Antibiotic treatment

SUMMARY:
In this randomized controlled trial the investigators want to compare the effect of one-time rectal instillation of fecal microbiota transplantation, compared to a ten-day antibiotic course for the treatment of primary Clostridium difficile infection (CDI). The investigators hypothetsize that the instillation of feces from a healthy donor will be non-inferior to vancomycin in inducing a durable cure.

DETAILED DESCRIPTION:
Up to one third of patients with clostridium difficile infection treated with antibiotics experience recurrent or relapsing symptoms within a few weeks. Even with subsequent antibiotic treatment, multiple recurrences/relapses are frequent. Fecal microbiota transplantation (FMT) has been shown to be significantly more effective in curing recurrent CDI than repeated antibiotic treatment. In current guidelines, FMT is proposed as a treatment option after multiple recurrences/relapses of CDI. The rationale to reserve transplantation of donor feces for recurrent and difficult cases of CDI is a possible risk of pathogen transmittance and the process of finding a donor and screen for communicable disease.

The effect of FMT for recurrent CDI, however, suggests that this therapy may be more effective than antibiotics in inducing a durable cure also for primary CDI. If the therapeutic effect of FMT proves to be equal (non-inferior) or more effective than antibiotics, FMT may be the preferable treatment option due to favourable ecological impact compared to antibiotics. In an era with increasing concerns about overuse of antibiotics and emergence of antibiotic resistant bacteria, it is important to investigate therapeutic alternatives that may reduce the need for antibiotics.

This trial is a phase III multicentre, randomized controlled, open-label non-inferiority parallel group trial with two arms (FMT and antibiotics), and is a continuation of the phase II trial IMT for Primary Clostridium Difficile Infection (NCT02301000). In the current trial, patients with Clostridium difficile infection and no previous CDI within 12 months prior to inclusion will be randomized 1:1 to FMT or 10 days of guideline-recommended antibiotic therapy (vancomycin 125 mg four times a day).

Patients are recruited in Norwegian hospitals.

The investigators plan to use frozen microbiota, because supply is easier to organize, compared to fresh fecal samples. Patients in the FMT treatment group will receive one rectal dose of FMT, originating from screened, healthy donors. Patients who are not cured by the first dose is offered a protocol defined additional FMT treatment. In the case of clinical deterioration, appropriate measures will be undertaken according to current guidelines.

Patient treatment outcomes are evaluated after 14, 60 and 365 days from inclusion and treatment initiation.

An interim analysis is planned after inclusion of the first 94 patients (corresponding to 50% of the planned number of patients).

ELIGIBILITY:
Inclusion Criteria:

* Patients, ≥18 years with primary C. difficile infection, defined by the following three criteria:

  1. Diarrhea as defined by the WHO (≥3 loose stools per day), and
  2. Positive stool test for toxin producing C. difficile, and
  3. No evidence of previous C. difficile infection during 365 days before enrolment.
* Written informed consent

Exclusion Criteria:

* Known presence of other stool pathogens known to cause diarrhea.
* Ongoing antibiotic treatment for other infections that cannot be stopped before study treatment administration.
* Inflammatory bowel disease or microscopic colitis.
* < 3 months life expectancy.
* Serious immunodeficiency, defined as one of the following:

  * Ongoing or recent chemotherapy and current or expected neutropenia with neutrophil count of < 500/μL.
  * Active severe immunocompromising disease.
* Inability to comply with protocol requirements.
* Need of intensive care.
* Known irritable bowel syndrome, diarrheal type.
* Pregnancy or nursing.
* Known or suspected toxic megacolon or ileus.
* Total or subtotal colectomy, ileostomy or colonostomy.
* Contraindications for rectal catheter insertion
* Known hypersensitivity or other contraindications to vancomycin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Patients with durable cure | 60 days
  Proportion of patients with primary clinical cure at day 14 after treatment start and no recurrent C. difficile infection during 60 days after treatment start, with the assigned treatment alone.

SECONDARY OUTCOMES:
Patients with durable cure with additional treatment. | 60 days
  Proportion of patients with primary clinical cure at day 14 after treatment start and no recurrent C. difficile infection during 60 days after treatment start, with or without the need of additional treatment (FMT, metronidazole or vancomycin).
Treatment adverse events | 60 and 365 days
  Proportion of patients with adverse events.
Patients with long-time cure | 365 days
  Proportion of patients with primary clinical cure at day 14 after treatment start and no recurrent C. difficile infection during 60 days after treatment start, and without recurrent C. difficile infection within 365 days after treatment start.
Health-economic evaluation | 365 days
  Health-economic analysis of the two compared treatment modalities

OTHER OUTCOMES:
Fecal composition and treatment outcome | 60 days
  Correlation in fecal composition changes before versus after treatment, and treatment outcome (such as bacterial diversity and fecal short chain fatty acids).
  Subgroup analyses will be performed for sex, age, co-morbidities, and FMT donor.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bretthauer, MD, PhD, Study Chair — Oslo Universitetssykehus HF, Rikshospitalet
Locations (18):
- Norway (18):
  - Vestre Viken HF, Bærum Hospital, Sandvika, Gjettum
  - Diakonhjemmet Hospital, Oslo, Oslo County
  - Ålesund Sjukehus, Ålesund
  - Haukeland universitetssykehus, Bergen
  - Nordlandssykehuset, Bodø
  - Sykehuset Østfold Kalnes, Grålum
  - UNN Harstad, Harstad
  - Sørlandet Hospital HF, Kristiansand
  - Sykehuset Levanger, Levanger
  - Sykehuset Innlandet HF, Lillehammer
  - Akershus University Hospital, Lørenskog
  - Lovisenberg sykehus, Oslo
  - Oslo University Hospital Rikshospitalet, Oslo
  - Oslo University Hospital Ullevål, Oslo
  - Telemark Hospital HF, Skien
  - Stavanger University Hospital, Stavanger
  - UNN Tromsø, Tromsø
  - Sykehuset i Vestfold, Tønsberg

IPD SHARING:
Plan to Share IPD: Undecided
The trial adheres to data sharing policies of the ICMJE. Data sharing is considered for each request by the principal investigators. Data sharing is not granted if they overlap with planned analyses. Data sharing requires all approvals by relevant authorities. Costs for data sharing will not be covered by the study group.

REFERENCES:
- [Background] McDonald LC, Gerding DN, Johnson S, Bakken JS, Carroll KC, Coffin SE, Dubberke ER, Garey KW, Gould CV, Kelly C, Loo V, Shaklee Sammons J, Sandora TJ, Wilcox MH. Clinical Practice Guidelines for Clostridium difficile Infection in Adults and Children: 2017 Update by the Infectious Diseases Society of America (IDSA) and Society for Healthcare Epidemiology of America (SHEA). Clin Infect Dis. 2018 Mar 19;66(7):987-994. doi: 10.1093/cid/ciy149. PMID 29562266
- [Background] Juul FE, Garborg K, Bretthauer M, Skudal H, Oines MN, Wiig H, Rose O, Seip B, Lamont JT, Midtvedt T, Valeur J, Kalager M, Holme O, Helsingen L, Loberg M, Adami HO. Fecal Microbiota Transplantation for Primary Clostridium difficile Infection. N Engl J Med. 2018 Jun 28;378(26):2535-2536. doi: 10.1056/NEJMc1803103. Epub 2018 Jun 2. No abstract available. PMID 29860912
- [Background] Leffler DA, Lamont JT. Clostridium difficile infection. N Engl J Med. 2015 Apr 16;372(16):1539-48. doi: 10.1056/NEJMra1403772. No abstract available. PMID 25875259
- [Background] van Nood E, Dijkgraaf MG, Keller JJ. Duodenal infusion of feces for recurrent Clostridium difficile. N Engl J Med. 2013 May 30;368(22):2145. doi: 10.1056/NEJMc1303919. No abstract available. PMID 23718168
- [Background] Kassam Z, Lee CH, Yuan Y, Hunt RH. Fecal microbiota transplantation for Clostridium difficile infection: systematic review and meta-analysis. Am J Gastroenterol. 2013 Apr;108(4):500-8. doi: 10.1038/ajg.2013.59. Epub 2013 Mar 19. PMID 23511459
- [Derived] Juul FE, Bretthauer M, Johnsen PH, Samy F, Tonby K, Berdal JE, Hoff DAL, Ofstad EH, Abraham A, Seip B, Wiig H, Rognstad OB, Glad IF, Valeur J, Nissen-Lie AE, Ness-Jensen E, Lund KMA, Skjevling LK, Hanevik K, Skudal H, Melsom EJ, Boyar R, Cooper TJ, Ranheim TE, Riise EM, Adami HO, Kalager M, Loberg M, Garborg KK. Fecal Microbiota Transplantation Versus Vancomycin for Primary Clostridioides difficile Infection : A Randomized Controlled Trial. Ann Intern Med. 2025 Jul;178(7):940-947. doi: 10.7326/ANNALS-24-03285. Epub 2025 Jun 17. PMID 40523286
- See also: Investigating research group' home page — https://www.med.uio.no/helsam/english/research/groups/clinical-effectiveness/index.html